CLINICAL TRIAL: NCT04479891
Title: A Single-centre, Open, Single-dose, Self-control Study to Investigate the Effect of Itraconazole on the Pharmacokinetics of Pyrotinib in Healthy Subjects
Brief Title: Effect of Itraconazole on the Pharmacokinetics of Pyrotinib in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HR-BLTN-DDI-01
Record Dates: First submitted 2020-07-17; First posted 2020-07-21 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — pyrotinib; Itraconazole

STUDY DESIGN:
Intervention Model Description: Pyrotinib alone and then combined with itraconazole
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pyrotinib alone, pyrotinib + itraconazole (Experimental): Sequential treatments of pyrotinib alone followed by pyrotinib + itraconazole, with a washout period in between.
  Interventions: Drug: pyrotinib tablet; Drug: Itraconazole capsule

INTERVENTIONS:
Drug: pyrotinib tablet — single oral dose of SHR6390 or co-administered with itraconazole
Drug: Itraconazole capsule — 200 mg itraconazole QD

SUMMARY:
The study will assess the effect of multiple oral doses of itraconazole on the single dose pharmacokinetic parameters of pyrotinib in healthy Chinese subjects. The safety of pyrotinib alone and when co-administered with itraconazole will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Sign the informed consent before the trial, and fully understand the trial content, process and possible adverse reactions;
* Able to complete the study as required by the protocol;
* Subjects have no birth plan and voluntarily take effective contraception from 2 weeks before administration to 3 months after the last dose, and the pre-drug serum HCG test for fertility-enabled women must be negative;
* Male body weight ≥ 50 kg, female body weight ≥ 45 kg, and body mass index (BMI) within the range of 19 ~ 26 kg/m2 ;
* No clinically significant abnormalities in general physical examination, vital signs, laboratory tests, etc.

Exclusion Criteria:

* Blood donation no less than 400 mL or have blood transfusion within 3 months of dosing.
* Allergic constitution or known allergy to pyrotinib, itraconazole or the excipients;
* History of drug abuse in the past 5 years, or positive for drug abuse screening;
* Alcoholic or often drinkers with drinking amount more than 14 units a week; a heavy smoker; and can't abstain from smoking and alcohol during the study
* Left ventricular ejection fraction (LVEF) <50% by echocardiography or QTcF ≥ 470 msec by 12 lead electrocardiograph;
* A clear medical history of important primary organ diseases such as nervous system, cardiovascular system, urinary system, digestive system, respiratory system, metabolism and musculoskeletal system that are not suitable for subjects to participate in the study, as judged by the investigator;
* Any surgery within 6 months before screening;
* Have taken hepatotoxic drugs for a long time within 6 months before screening;
* Subjects who took any clinical trial drugs within 3 months;
* Subjects who took any drugs that change liver enzymes activity within 28 days before dosing; or took any prescription drugs, over-the-counter drugs or vitamins, health products or herbal medicine within 14 days before dosing;
* Hepatitis B surface antigen positive, hepatitis C antibody positive, syphilis antibody positive, HIV antibody positive;
* Subjects who took any beverage or food containing grapefruit, xanthine, caffeine, or alcohol within 48 hours before dosing; strenuous exercise; or other factors which affect drug absorption, distribution, metabolism, excretion, etc.;
* Other factors that are not suitable for subjects to participate in the study, as judged by the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2019-09-18 (Actual); Primary Completion 2019-10-11 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Cmax of pyrotinib | Day 1 and Day 9
  Maximum concentration (Cmax) of pyrotinib
AUC of pyrotinib | Day 1 and Day 9
  Area under the plasma concentration versus time curve of SHR6390

SECONDARY OUTCOMES:
Tmax of pyrotinib | Day 1 and Day 9
  Time of maximum concentration of pyrotinib
T1/2 of pyrotinib | Day 1 and Day 9
  Terminal half-life of pyrotinib
AEs and SAEs | From the first drug administration to 7 days after the last drug administration
  Adverse events and serious adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital of Anhui Medical University, Hefei, Anhui, China